CLINICAL TRIAL: NCT01612728
Title: Aromatase Inhibitor-Induced Arthralgia: A Proposed Management Algorithm
Brief Title: Treatment for Joint Pains Due to Aromatase Inhibitor Therapy in Breast Cancer
Acronym: AIA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The grant application for this project was rejected.
Sponsor: Baylor Breast Care Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIA-001
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer; Arthralgia; Joint Pain
Keywords: Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women with Arthralgia (Experimental): Women who develop joint pain on Aromatase Inhibitor therapy will be placed on the clinical algorithm, as specified in the protocol.
  Interventions: Drug: Women with Arthralgia
- Women without Arthralgia (Other): Women who do not develop arthralgia will continue to have their joint pain and strength measured, as well as their medication compliance. However, they will not be placed on the clinical algorithm which is meant for alleviation of joint pains.
  Interventions: Other: Women without Arthralgia

INTERVENTIONS:
Other: Women without Arthralgia — For mild arthralgia, women will try the following interventions in the following order: 1) Weight-bearing exercise program, and 2) Glucosamine & Chondroitin supplements. For women with mild to moderate arthralgia, they will try to the following interventions in this order: 1) Acupuncture, 2) Indomethacin twice daily as needed, 3) Switch to a different aromatase inhibitor, and 4) Switch to tamoxifen.
  Arms: Women without Arthralgia
Drug: Women with Arthralgia
  Other Names: Aromatase Inhibitor
  Arms: Women with Arthralgia

SUMMARY:
Aromatase inhibitors are the most effective adjuvant anti-hormonal therapy for estrogen receptor positive (ER+) post-menopausal breast cancer patients, with proven superiority over tamoxifen in terms of disease-free survival, time to recurrence, and contralateral breast cancer. However, approximately half of the women who take this drug will develop significant joint pains, termed Aromatase Inhibitor-Induced Arthralgia (AIA). Though this medicine should be taken for 5 years, the joint pain can be so troublesome that up to 13% may prematurely discontinue it because of the arthralgia, thus sacrificing their best chance of recurrence-free survival. Nonetheless, neither the etiology nor optimal management of AIA is clearly understood, leaving both doctor and patient rather frustrated.

The investigators therefore propose to test the hypothesis that AIA can be effectively treated by a new clinical algorithm, and that effective treatment of the problem will lead to improved compliance with Aromatase Inhibitor (AI) therapy. The algorithm is a clinical pathway for treating AIA which incorporates, in a rational and step-wise manner, a series of interventions based on the available evidence. Interventions include acupuncture, pain medication, weight bearing exercise, and other commonly used therapies for AIA.

The investigators will enroll 100 women who are beginning adjuvant AI therapy and assess each woman's baseline joint pains via a questionnaire as well as grip strength measurement. The investigators will then periodically repeat these tests during AI therapy in order to systematically quantify and characterize AIA. Those women who develop AIA during the course of the study will be placed on the clinical algorithm, and the investigators will observe whether their joint pains significantly improve (as measured by questionnaire and grip strength measurement) after institution of the algorithm. The investigators will also determine whether their compliance is improved compared to historical controls, and at least non-inferior to the women in the study who do not develop AIA. Finally, the investigators will measure serum estrogen level at baseline and then periodically during AI therapy to investigate whether more dramatic decline in estrogen level after initiation of an AI leads to significant AIA and earlier time to onset.

This study targets a very common cause of pain among breast cancer survivors and aims to offer an effective treatment strategy to alleviate pain and improve quality of life as well as medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* stage I-III ER+ breast cancer
* beginning adjuvant AI therapy
* post-menopausal as defined by any of the following: age >60 years, history of bilateral oophorectomy, amenorrhea for 1 year with intact uterus and ovaries, or serum estradiol and FSH concentrations in the post-menopausal range along with either amenorrhea for 6 months or previous hysterectomy

Exclusion Criteria:

* previous use of an aromatase inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Medication compliance | 9 months
  The primary objective of the study will be to estimate medication compliance among women with and without arthralgia with use of the proposed algorithm in those women with AIA.

SECONDARY OUTCOMES:
improvement of AIA symptoms with use of the algorithm | 9 months
  The secondary objectives of the study will be correlation of the estrogen level with clinical development of arthralgia, as well as greater improvement of AIA symptoms with use of the algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Niravath, MD, Principal Investigator — Baylor College of Medicine